CLINICAL TRIAL: NCT03852888
Title: Kinetics of Elimination of Methotrexate and Its Major Metabolite 7-OH-methotrexate for Observant Patients
Acronym: MetU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PO18172*
Record Dates: First submitted 2019-02-07; First posted 2019-02-25 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2021-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mtugroup (Experimental): All patients managed for rheumatoid arthritis (according to the ACR / EULAR 2010 criteria) in the Rheumatology Department of the University Hospital of Reims and treated with methotrexate monotherapy.
  Interventions: Biological: Urine samples taken to measure methotrexate and its major metabolite 7-OH-methotrexate level

INTERVENTIONS:
Biological: Urine samples taken to measure methotrexate and its major metabolite 7-OH-methotrexate level — Each patient will have to complete a total of 8 urine samples after treatment with methotrexate. The 8 samples will be taken over one week (just before taking, then 2 hours after taking treatment and then on D3, D4, D5, D6, D7, D8 before the new dose of methotrexate).

SUMMARY:
Methotrexate is a key treatment for inflammatory rheumatism. Therapeutic compliance with methotrexate is difficult to measure because of a lack of objective testing; however, therapeutic compliance is essential for the proper management of a patient.

The objective is to characterize the kinetics of elimination of methotrexate and its main metabolite7-OH-methotrexate for observant patients according to treatment (dosage, administration) and patient characteristics.

Once this kinetics is characterized, it will be considered as a comparison reference to identify non-observant patients that is to say having concentrations lower than the lower bound of the confidence interval of the observed concentrations.

DETAILED DESCRIPTION:
Type of study: prospective longitudinal descriptive observational study Population: Patients treated for rheumatoid arthritis in the Rheumatology Department of Reims University Hospital and treated with methotrexate monotherapy (weekly intake).

Assessment Criteria: Urinary concentration of methotrexate and its metabolite 7-OH-methotrexate at different days post-administration.

Investigation plan: Determination of urinary methotrexate and its 7-OH-methotrexate metabolite on 8 urine samples (just before taking, then 2 hours after treatment and then on D3, D4, D5, D6, D7, D8 before re-taking methotrexate) in the same patient treated with methotrexate weekly. It will take 10 patients per dosage level, followed by 3 to 8 days post-administration, to distinguish the urinary methotrexate concentrations of observant patients from those of non-observant patients with the power of 90%.

Statistical Analysis Plan: The main objective of this study is to characterize the elimination kinetics of methotrexate and its major metabolite 7-OH-methotrexate in patients observing the various methotrexate regimens. Once this kinetics is characterized, it will be considered as a comparison reference to identify non-observant patients that is to say having concentrations lower than the lower bound of the confidence interval of the observed concentrations.

On the one hand, simulations based on published population pharmacokinetic models of plasma methotrexate are used to estimate the periods of elimination of methotrexate. The simulations that the investigators carried out on the basis of these models highlight that these elimination periods are between 3 and at the latest 9.5 days. These periods correspond to the time required to eliminate 99% of methotrexate.

Finally, it will take 10 patients per dosage level, by administration (oral or subcutaneous), followed by the 3rd to 8th day post-administration, to distinguish urinary methotrexate concentrations from observant patients (1 +/- 0.3 nM) of non-observant patients (0.4 +/- 0.4 nM) with the power of 90%. The dosage schedules are 10, 15, 20 mg methotrexate / week per-os or subcutaneous injection. It will recruit 60 patients. The follow-up will be limited to 8 days maximum because the administration is done once a week.

ELIGIBILITY:
Inclusion Criteria:

* All patients managed for rheumatoid arthritis (according to the ACR / EULAR 2010 criteria) in the Rheumatology Department of the University Hospital of Reims and treated with methotrexate monotherapy.
* Patient affiliated to a social security scheme.

Exclusion Criteria:

* Patient protected by law.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2021-11-25 (Actual)

PRIMARY OUTCOMES:
Urinary concentration of methotrexate and its major metabolite 7-OH-methotrexate | Day 8
  LC-MS/MS quantification (in nM)

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Theate N, Geoffroy M, Kanagaratnam L, Gozalo C, Charlot I, Bolko L, Hittinger-Roux A, Djerada Z, Salmon JH. Urinary methotrexate dosage in rheumatoid arthritis, in patients treated for at least 6 months: a potential marker of adherence. RMD Open. 2024 May 20;10(2):e004024. doi: 10.1136/rmdopen-2023-004024. PMID 38772677